CLINICAL TRIAL: NCT00284063
Title: Z-Joint Changes in Low Back Pain Following Adjusting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Health Sciences (Other)
Collaborators: Canadian Memorial Chiropractic College (Other); Auburn University (Other)
Responsible Party: Principal Investigator, Gregory D. Cramer, Dean of Research, National University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2R01AT000123-03 (NIH)
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2022-05-12 (Actual); Status verified 2015-04

CONDITIONS: Mechanical Low Back Pain
Keywords: spinal manipulation, zygapophysial joints
MeSH Terms: conditions — Low Back Pain | interventions — Magnetic Resonance Spectroscopy; Manipulation, Chiropractic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1: N; SPP; N (Active Comparator): N = neutral MRI; SP = side posture MRI; SPP = side posture position; SMT = side posture manipulation
  Interventions: Procedure: MRI
- Group 2: N; SMT; N (Active Comparator): N = neutral MRI; SP = side posture MRI; SPP = side posture position; SMT = side posture manipulation
  Interventions: Procedure: Low back adjustment and MRI
- Group 3: N; SMT; SP (Active Comparator): N = neutral MRI; SP = side posture MRI; SPP = side posture position; SMT = side posture manipulation
  Interventions: Procedure: Low back adjustment and MRI
- Group 4: N and SP (No Intervention): N = neutral MRI SP = side posture MRI SPP = side posture position SMT = side posture manipulation

INTERVENTIONS:
Procedure: Low back adjustment and MRI — Subjects received a 15 minutes MRI in neutral position, a chiropractic low back spinal manipulation, and a second 15 minute MRI in neutral position.
  Other Names: spinal manipulation = spinal adjustment
  Arms: Group 2: N; SMT; N
Procedure: Low back adjustment and MRI — Subjects received a 15 minutes MRI in neutral position, a chiropractic spinal manipulation to the low back, and a second 15 minute MRI in a side posture position.
  Other Names: spinal manipulation = spinal adjustment
  Arms: Group 3: N; SMT; SP
Procedure: MRI — Subjects received a 15 minute MRI in neutral position and a second 15 minute MRI in neutral position.
  Other Names: spinal manipulation = spinal adjustment
  Arms: Group 1: N; SPP; N

SUMMARY:
The purpose of this continuation project is to use MRI to evaluate gapping of the zygapophysial (Z) joints following side-posture positioning and side-posture spinal adjusting in subjects with acute low back pain.

DETAILED DESCRIPTION:
The purpose of this continuation project is to use MRI to evaluate gapping of the zygapophysial (Z) joints following side-posture positioning and side-posture spinal adjusting in subjects with acute low back pain (LBP). A fundamental hypothesis of one of the beneficial effects of chiropractic spinal adjusting is that adhesions, developing in the Z joints following hypomobility of these structures, are thought to be alleviated by separation (gapping) of the Z joints through spinal adjusting. In the previous study, side-posture adjusting was found to gap the Z joints in healthy subjects. The aim of this study is to determine if differences can be measured in the L4/L5 and L5/S1 Z joint spaces during side-posture positioning and after lumbar side-posture spinal adjusting of 112 subjects with acute LBP, and to determine if the amount of gapping is related to pain relief and improved function. Before any treatment begins, the subjects will be temporarily randomized into one of 4 MRI groups: 1) neutral positioning, followed by side-posture positioning (most painful side up); 2) neutral positioning, followed by side-posture adjusting (most painful side up), followed by neutral positioning; 3) neutral positioning, followed by side-posture adjusting (most painful side up) and remaining in side-posture; and 4) (pure control group) neutral positioning, followed by very brief side-posture positioning, followed by neutral positioning. MRI scans will be taken with the subjects in the original neutral position and in the final position. Both MRI scans will be conducted consecutively over approximately 30 minutes (12:19 minutes per scan). All spinal adjustments given during this appointment will be performed directly on the MRI gantry table after the first scan. A second MRI appointment will occur 2 weeks later, after 2 weeks of treatment. At the second MRI appointment, subjects will be assigned to the MRI group opposite to the one to which they were randomized during the first MRI appointment. Three observers, blinded to each other and to subject grouping, will make anterior-to-posterior measurements (A-P gap) of the Z joints directly from the MRI scans. The gapping difference between the second and first scans of each MRI appointment will be analyzed to determine if differences exist between the 4 groups. Results of the first and second MRI appointments will also be evaluated to determine if the amount of gapping is related to pain (at first MRI appointment), relief of pain (at the second MRI appointment - difference in Visual Analog Scale from initial exam to MRI appointment) and current (first MRI appointment) and change in disability (second MRI appointment - difference in Bournemouth Questionnaire scores). The results of this study will be used to increase understanding of the mechanism of action of lumbar side posture adjusting and side-posture positioning in acute LBP patients.

ELIGIBILITY:
Inclusion Criteria:

* Twenty-one to 69 years of age (21 years to ensure fully developed Z joints and <70 years to tolerate side posture MRI scans)
* Females equal to or less than 160 pounds; males equal to or less than 200 pounds. Hip width measurement that is equal to or less than 36cm.(to ensure optimum MR image quality)
* Pain related to the low back (lower lumbar region, L4/L5 and/or L5/S1 region -this criterion will be determined by the examining physician through subjective complaint and description, as well as objectively, using inspection, palpation, motion assessment, and standard orthopedic and neurologic tests
* No history of LBP lasting for more than two weeks, or no more than 3 episodes of brief back pain (1 - 2 weeks) in the past year.

Exclusion Criteria:

* Presence of lumbar scoliosis of greater than 5 degrees (Cobb's angle) (due to difficulty in imaging the Z joints)
* Presence of radiculopathy (This criterion will be evaluated by the examining physician by using patient history, standard screening tests, and the results of a detailed orthopedic/neurologic evaluation).
* No pain related to L4/L5 and/or L5/S1 region (This criterion will be determined by the examining physician through subjective complaint and description, as well as objectively using inspection, palpation, motion assessment, and standard orthopedic tests such as, Kemp's, Milgram's, Yeoman's, straight leg raise, and Valsalva maneuver.)
* Pregnancy or currently breast feeding (for MRI, even though no known risk, and in the event an x-ray is needed to screen for contraindications to manipulation)
* Intolerance to MRI procedures (including claustrophobia and inability to lie on one's side for 15 minutes). This criterion can also be evaluated at any time throughout the first two weeks of a subject's care. Claustrophobia will also be evaluated before and during the first and second MRI scans.
* Significant pathology discovered on MRI scans. This criterion will be evaluated during the first MRI visit, immediately after the first MRI scan is taken. (Such pathologies constitute contraindications to chiropractic adjusting.)
* Absence of acute low back pain

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2006-01-31 (Actual); Primary Completion 2009-12-01 (Actual); Study Completion 2010-09-30 (Actual)

PRIMARY OUTCOMES:
Anterior to posterior measurements (A-P gap) of the Z joints. | February 2006-December 2011

SECONDARY OUTCOMES:
Amount of gapping will be compared to relief of pain (Visual Analog Scale). | February 2006-January 2010
Amount of gapping compared to disability (Bournemouth Questionnaire) | February 2006-January 2009

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D. Cramer, DC, PhD, Principal Investigator — National University of Health Sciences
Locations (1):
- National University of Health Sciences, Lombard, Illinois, United States